CLINICAL TRIAL: NCT01491061
Title: TWice overnIght High-dose ranoLazIne Pretreatment for preventinG Myocardial iscHemic Damage in Patients With Stable Angina Undergoing percuTaneous Coronary Intervention
Brief Title: Ranolazine Loading to Prevent PCI-induced Myocardial Injury
Acronym: TWILIGHT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 653/2011/D
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: periprocedural myocardial infarction; ranolazine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): Administration of two preprocedural doses of Ranolazine 12 hours apart (1,000 mg the night before PCI and 1,000 mg prior to PCI)
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — os, 1,000 mg twice 12 hours apart prior to PCI
  Other Names: Ranexa TM, Gilead, USA
  Arms: Ranolazine
Drug: Placebo — os, two doses 12 hours apart prior to PCI
  Arms: Placebo

SUMMARY:
It has previously been shown that pretreatment with ranolazine 1,000 mg twice daily for 7 days can significantly reduce procedural myocardial injury in elective percutaneous coronary intervention (PCI). The investigators tested the hypothesis that twice overnight high-dose ranolazine loading before PCI can reduce the peri-procedural myocardial ischemic damage similarly to long-term pre-treatment with standard doses.

DETAILED DESCRIPTION:
Background

Ranolazine is a novel antianginal drug that reduces intracellular sodium and calcium accumulation during ischemia thus limiting ischemic injury.

It has previously been shown that pretreatment with ranolazine 1,000 mg twice daily for 7 days can significantly reduce procedural myocardial injury in elective percutaneous coronary intervention.

It remains unknown, however, which of these two therapeutic approaches is more effective after PCI.

Purpose

The primary objective of this study is to test the hypothesis that twice overnight high-dose ranolazine loading before PCI can reduce the peri-procedural myocardial ischemic damage similarly to long-term pre-treatment with standard doses.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Class I indication to elective percutaneous coronary intervention
* Stable conditions
* No recent acute coronary syndromes
* Normal baseline values of markers of myocardial damage (creatine kinase, creatine kinase-MB, myoglobin, and troponin I)
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of PCI-induced myocardial infarction | Up to 48 hours after PCI
  Occurrence of peri-procedural myocardial infarction (i.e. creatine kinase-MB>3 times the upper reference limit)

SECONDARY OUTCOMES:
Assessment of post-PCI peak values of markers of myocardial damage | Baseline and 48 hours after PCI
  Changes after percutaneous coronary intervention in absolute values of creatine kinase, creatine kinase-MB, myoglobin, and troponin I
Rate of 30-day MACE | Up to 30 days after PCI
  30-day incidence of major adverse cardiac events (MACE-death, myocardial infarction, target vessel revascularization)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Pisana, Rome, Italy